CLINICAL TRIAL: NCT05939960
Title: Application of a New Type of Whole Blood Coagulation Time Measurement in Evaluating the Hypercoagulable State of Malignant Tumors
Acronym: GCTHCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qiong Qin, Director of Oncology Department, Tianjin Medical University General Hospital
Other Study IDs: IRB2023-RTFL-134
Record Dates: First submitted 2023-07-01; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Neoplasm Metastasis; Blood Coagulation Disorder With Shortened Coagulation Time (Disorder); Venous Thromboembolism
Keywords: Neoplasm Metastasis; Blood Coagulation Disorder; Venous Thromboembolism
MeSH Terms: conditions — Neoplasm Metastasis; Venous Thromboembolism; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal group: GCT time within normal range；Normal coagulation function
  Interventions: Diagnostic Test: CGT test
- hypercoagulable group: GCT time reduction； Normal coagulation function,
  Interventions: Diagnostic Test: CGT test

INTERVENTIONS:
Diagnostic Test: CGT test — GCT、PRP-CT、PPP-CT monitor

SUMMARY:
Malignant tumors are closely related to deep vein thrombosis, Pulmonary embolism and other diseases. Tumor patients usually have a hypercoagulable state (HCS) in their blood, and the proportion of thrombosis caused by HCS is more than 10 times that of non tumor patients. Conventional clinical testing methods such as coagulation function, blood routine, and thromboelastography are difficult to directly evaluate the hypercoagulable state of tumor patients. In addition, the widely used Khorana score and Caprini score systems in clinical practice need to be improved in accurately reflecting the hypercoagulable state of tumor patients.

Our team has established a complete new coagulation time measurement system, including general clotting time (GCT), platelet rich plasma clotting time (PRP-CT), and platelet poor plasma clotting time (PPP-CT), which may be a new and accurate method for evaluating tumor hypercoagulability.

The GCT study aims to evaluate: 1. The time of GCT, PRP-CT, and PPP-CT for malignant tumors is shorter than that of normal individuals, and some patients are in a hypercoagulable state; 2. The shortened time of GCT, PRP-CT, and PPP-CT may be associated with future thrombosis; 3. Evaluating the relationship between shortened GCT system time and overall tumor survival

Therefore, the GCT system evaluation may identify patients who are truly in a hypercoagulable state, providing monitoring indicators for subsequent anticoagulation; It can also be evaluated whether GCT time can reflect the prognosis of tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign an informed consent form;
2. Age ≥ 18 years old
3. Expected survival time>6 months;
4. Patients diagnosed with malignant tumors for the first time or progressing during treatment;
5. Solid malignant tumors with clear pathological diagnosis;
6. ECOG physical fitness score ≤ 2 points

Exclusion Criteria:

1. Patients with known venous thrombosis (including upper and lower limb venous thrombosis, Pulmonary embolism, visceral venous thrombosis, etc.);
2. Patients who have received long-term treatment with Warfarin, Rivaroxaban, and low-molecular-weight heparin (except aspirin, hydrogen Clopidogrel, etc.);
3. Patients with active infections and sepsis;
4. Hematology tumor (except lymphoma);
5. Patients who undergo any major surgical treatment within 28 days prior to enrollment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the commonly used Caprini Thrombosis Risk Score and Khrona Thrombosis Risk Score in clinical practice, patients with Caprini score ≥ 5 and Khrona score ≥ 2 have a VTE incidence rate of 8.8% -14.6%; The expected incidence of VTE in patients with shortened whole blood GCT time is 30%; Based on sample size calculation, Class I error α= 0.025, Class II error β= 0.05, bilateral test, loss of follow-up rate of 10%, calculated sample size of 76 cases. It is predicted that patients with shortened GCT time account for 30% of all tumor patients, and 254 patients need to complete GCT testing. Therefore, the overall sample size required for this study is 254 cases.
Sampling Method: Probability Sample
Enrollment: 354 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Compared with non tumor patients, the GCT time of tumor patients is significantly GCT shortened in neoplames | July 1,2023 to September 30,2024
  Compared with non tumor patients, the GCT time of tumor patients is significantly shortened

SECONDARY OUTCOMES:
theincreased incidence of VTE | July 1,2023 to September 30,2024
  In patients with shortened GCT, the incidence of VTE increases.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jianning, Doctor, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
After completing the research thoroughly, apply for and obtain the consent of PI to access the data